CLINICAL TRIAL: NCT02570230
Title: Low Dose Intraoperative Intravenous Ketamine Combination With Spinal Morphine for Post Thoracic Surgery Pain : A Randomized Control Study
Brief Title: Ketamine Combination With Spinal Morphine for Post Thoracic Surgery Pain : A Randomized Control Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI2558
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Pain; Postoperative Period
Keywords: Thoracotomy; Postoperative pain; Ketamine
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): NSS infusion
  Interventions: Other: NSS
- Ketamine (Experimental): Ketamine 0.2 mg/kg/hr intravenous infusion
  Interventions: Drug: Ketamine

INTERVENTIONS:
Other: NSS — NSS infusion
  Arms: Control
Drug: Ketamine — Ketamine 0.2 mg/kg/hr intravenous infusion
  Arms: Ketamine

SUMMARY:
Thoracotomy is one of the most painful operation. Continuous thoracic epidural or paravertebral analgesia are gold standard for postoperative pain. But both techniques require skills. Spinal morphine is alternative simple method with less efficacy. Adding low dose ketamine during intraoperative may be helpful in postoperative pain relief.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3
* elective thoracotomy
* can operate patient-controlled analgesia (PCA) machine

Exclusion Criteria:

patient with history of

* allergy to morphine or ketamine
* contraindicate to ketamine
* remain intubated in the postoperative period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Time to first trigger of morphine | 24 hours
  Time to first trigger of morphine

SECONDARY OUTCOMES:
24-hr morphine consumption | 24 hours
  24-hr morphine consumption
NRS score at 6, 24 hours | 24 hours
  NRS score (0-10) was assessed at at 6, 24 hours postoperative
Incidence of nausea and vomiting | 24 hours
  Incidence of nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No